CLINICAL TRIAL: NCT03805048
Title: PeRcutaneous cOronary Intervention of Native Coronary arTery Versus Venous Bypass Graft in Patients With Prior cORonary Artery Bypass Graft Surgery - the PROCTOR Trial
Brief Title: PeRcutaneous cOronary Intervention of Native Coronary arTery Versus Venous Bypass Graft in Patients With Prior CABG
Acronym: PROCTOR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Paul Knaapen, Prinicipal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amsterdam UMC
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Dysfunctional venous bypass graft; Second generation DES; CABG
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either native vessel PCI or PCI of the venous bypass graft in a 1:1 fashion. Randomization will be performed using an interactive Web-based randomization system, Open Clinica
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Native Vessel PCI (Other): All patients with a significant stenosis (>50% on coronary angiography) in a venous bypass graft discussed in the local heart team for revascularization will be screened for potential inclusion in the study. Percutaneous coronary intervention of the native vessel will be performed according to current standard. In case of a CTO lesion, the aforementioned hybrid approach will be applied.This approach uses several angiographic characteristics to guide strategical planning of the procedure, using four complementary techniques to cross a CTO: antegrade wire escalation, antegrade dissection reentry, retrograde wire escalation and retrograde dissection reentry.
  Interventions: Procedure: Percutaneous coronary intervention
- Graft PCI (Other): All patients with a significant stenosis (>50% on coronary angiography) in a venous bypass graft discussed in the local heart team for revascularization will be screened for potential inclusion in the study. Percutaneous coronary intervention of the bypass graft will be performed following current standards and at the discretion of the operating interventional cardiologist. Only commercially available second generation DES will be used in the treatment of bypass grafts. The second generation DES used in this study will be the XIENCE Sierra stent. The use of a filter-wire during the procedure will be left at the discretion of the operator.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — PCI of the bypass graft will be performed by current standards and at the discretion of the operator. Only commercially available second generation DES - XIENCE Sierra will be used. In case of a CTO lesion, the aforementioned hybrid approach will be applied.This approach uses several angiographic characteristics to guide strategical planning of the procedure, using 4 complementary techniques to cross a CTO: antegrade wire escalation, antegrade dissection reentry, retrograde wire escalation, retrograde dissection reentry. In case of PCI failure, a second attempt can be performed within 1 month. Patients will be hospitalized for a min. of 6-8 hours after PCI and receive DAPT prior to the procedure or triple therapy in case of indication for oral anticoagulation, their duration according to the current guidelines of the ESC for stable coronary disease or ACS.

SUMMARY:
Multi-centre, randomised clinical trial with anticipated 17 European centres: in the Netherlands, Belgium, Germany and UK. Patients with a dysfunctional bypass graft with a clinical indication for revascularization will be randomized to either PCI of the native vessel or PCI of the dysfunctional venous bypass graft. 584 patients with a a clinical indication for percutaneous coronary intervention and a dysfunctional graft on the target vesselional venous bypass graft are planned to be enrolled during 3 years.Study objectives: to investigate the clinical and angiographic outcome of native vessel PCI compared to PCI of venous bypass graft in patients with a dysfunctional venous bypass graft with a clinical indication for revascularization. 1 year and 5 years, follow-up will be performed by means of a telephonic visit. After 3 years patients will be admitted to undergo a control invasive angiography.The CT-substudy and the PROCTOR registry is planned to be conducted too.

DETAILED DESCRIPTION:
Multi-centre, randomised clinical trial with anticipated 17 European centres: in the Netherlands, Belgium, Germany and UK. Patients with a dysfunctional bypass graft with a clinical indication for revascularization will be randomized to either PCI of the native vessel or PCI of the dysfunctional venous bypass graft. The CT-substudy and the PROCTOR registry is planned to be conducted too (details included in the flow chart).

CCTA substudy Selected patients will be approached for participation in the CCTA substudy of the trial. Participation in this substudy is optional. After written informed consent is obtained patients will undergo a CCTA in an out-patient setting. The CCTA will be performed before the PCI procedure.

PROCTOR registry

Patients can be approached for the registry when :

* PCI have been deemed clinically indicated by the local hartteam, and
* both the lesions in the native vessel and the dysfunctional graft have been deemed technically feasible by the local hartteam,
* the patient does not meet the in- and exclusion criteria for the randomized PROCTOR study or declines to participate in the randomized study.

Patients will be approached for participation and will have one week to consider. Written informed consent is mandatory for participating in the registry. Patients will be followed by telephonic follow-up after 1, 3, and 5 years. No additional study procedures will be performed.

Study objectives:to investigate the clinical and angiographic outcome of native vessel PCI compared to PCI of venous bypass graft in patients with a dysfunctional venous bypass graft with a clinical indication for revascularization.

1. PROCTOR main study

   - Investigate the clinical outcome of native vessel PCI vs. PCI of dysfunctional venous bypass graft with a clinical indication for revascularisation
2. CCTA substudy

   * Investigate prognostic value of CT-derived plaque characteristics for occurrence of MACE following bypass graft PCI
   * Investigate value of CCTA in guidance of CTO PCI procedures
3. PROCTOR Registry - Investigate long-term clinical outcomes in patients with dysfunctional venous bypass graft and an indication for PCI whom are not included in randomised main study.

All patients with a significant stenosis (>50% on coronary angiography) in a venous bypass graft discussed in the local heart team for revascularization will be screened for potential inclusion in the study. Patients will be eligible for inclusion if revascularization is deemed clinically indicated and technically feasible for PCI by the local heart team. The indication for revascularization will be based on symptoms and evidence of ischemia and viability in the target vessel territory. The lesion in the native vessel must be bypassed by a single venous graft or must be connected to a jump graft at the most distal anastomosis of that graft. In jump grafts, the lesion must be located distally to the second-to-last anastomosis. In case both the lesion in the native vessel and the lesion in the graft are deemed technically feasible for PCI, patients will be eligible for inclusion in the randomized study after consideration of in- and exclusion criteria. Patients who do not meet these criteria or decline to participate in the randomized study will be approached for inclusion in the registry. Subsequently patients will be approached for study participation. After being informed, patients will have at least 24 hours to consider participation. An independent physician will be available for extra information, if desired. After obtaining written informed consent, patients will be randomized to either native vessel PCI or PCI of the venous bypass graft. In case of PCI failure, a second attempt can be performed by the operator within one month.

If feasible, it is possible to perform a second attempt in another high-volume center. When successful PCI cannot be accomplished in one or two attempts, cross-over to the other treatment arm may be used as bailout strategy to restore myocardial blood flow to the distal vascular bed of the vessel. Randomization will be performed using an interactive Web-based randomization system, Open Clinica. After 1 and 5 years, follow-up will be performed by means of a telephonic visit. After 3 years patients will be admitted to undergo a control invasive angiography.

ELIGIBILITY:
Inclusion Criteria:

* A significant stenosis (>50% on angiography) in a venous bypass graft

  * The native lesion must be bypassed by a single graft or must be connected to a jump graft at the most distal anastomosis of that graft
  * In jumpgraft lesions, the lesion must be located distally to the second-to-last anastomosis
* Clinical indication for revascularization as determined by the local heart team (based on symptoms, documented ischemia, and viability).
* Both the native lesion and the venous graft lesion must be deemed suitable for PCI with a commercially available second generation DES.
* Informed consent must be obtained

Exclusion Criteria:

* < 18 years of age
* Target vessel diameter < 2.5 mm
* CABG performed less than 1 year prior to inclusion
* Diameter of the graft > 5.5 mm
* Aneurysm formation in the bypass graft
* Heavy burden of thrombus in the bypass graft (>50% of the bypass graft lumen in ≥2 out of 3 of the proximal, middle or distal third of the bypass graft).
* STEMI at presentation
* NSTEMI patients with ongoing ischemia
* Cardiogenic shock
* Severe kidney disease defined as an eGFR < 30 ml/min.
* Pregnancy
* Estimated life expectancy < 3 year
* Contraindications to PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Amount and type of Major Adverse Cardiac Events | 3 year follow up
  The total number and specification of major adverse cardiac events (all-cause mortality, non-fatal myocardial infarction, or clinically driven target lesion revascularization).

SECONDARY OUTCOMES:
Amount and type of Major Adverse Cardiac Events | 1 and 5 year follow-up
  The total number and specification of major adverse cardiac events (all-cause mortality, non-fatal myocardial infarction, or clinically driven target lesion revascularization).
Amount of patients that have passed away | 1, 3 and 5 year follow-up
  Mortality score, all-cause mortality
Number of non-fatal myocardial infarctions | 1, 3 and 5 year follow-up
  Any non-fatal myocardial infarction noticed
Number of clinically driven target lesion revascularizations | 1, 3 and 5 year follow-up
  Any clinically driven target lesion revascularization noticed
Number of target vessel revascularizations | 1, 3 and 5 year follow-up
  Any target vessel revascularization noticed.
Number of target vessel failure. | 1, 3 and 5 year follow-up
  Any target vessel failure noticed
Number of non-fatal myocardial infarctions. | >48 hours after PCI
  Any non-fatal myocardial infarction noticed.
Number of PCI-related myocardial infarctions. | 1, 3 and 5 year follow-up
  Any PCI-related myocardial infarction noticed.
Specific angiographic outcome | 3-year follow up
  Any of the following outcomes:
  * Late lumen loss
  * In-stent binary restenosis (≥50%)
  * In-stent re-occlusion
  * Difference in in-stent diameter stenosis between index procedure at inclusion, and at 3-year follow-up
Quality of life assessed by SAQ | 1, 3 and 5 year follow-up
  The Seattle Angina Questionnaire is a self-assessment questionnaire where patients' physical limitations caused by angina are quantified, as well as the frequency of and changes in their symptoms, their satisfaction with treatment and how they perceive their Quality of Life. Each scale is transformed to a 0-100 scale. the higher the score, the better the patients functions/the higher the Quality of Life.
Quality of life assessed by CCS | 1, 3 and 5 year follow-up
  Canadian Cardiovascular Society (CCS) Grading Scale measures whether patient have angina pectoris complaints, and to what extent patients experienced this. It uses a scale of 1-4 where 1 means angina pectoris (chest pain) only occurs with streneous, rapid or prolonged exertion, and 4 means angina is present during little physical effort or even during rest.
Quality of life assessed by RDS | 1, 3 and 5 year follow-up
  Rose dyspnea scale questionnaire (RDS) measures dyspnea complaints, or shortness of breath. It consists of 4 questions about dysnpea complaints in the everyday life of patients. For every patient, a score is compiled of the highest limitation in daily life, resulting in a score of 0-4, where 0 means no dyspnea complaints and 4 means the patient has complaints during no or minimal physical effort.
  The scores from these questionnaires will be combined by summing the total scores.
Composite score of quality of life | 3-year follow-up
  Composite of all quality of life questionnaires, where all outcomes are summed to provide a total score

CONTACTS AND LOCATIONS:
Overall Officials: Paul Knaapen, Principal Investigator — Amsterdam UMC
Locations (21):
- Belgium (4):
  - University Hospital, Antwerp, Edegem
  - Ziekenhuis Netwerk Antwerpen (ZNA) Middelheim, Antwerp
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Leuven, Leuven
- Universitäts Herzzentrum, Bad Krozingen, Germany
- Netherlands (8):
  - Universitair Medische Centra, Amsterdam
  - Academic Medical Center, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Radboud Universitair Medisch Centrum (Radboud UMC), Nijmegen
  - Universitair Medisch Centrum, Utrecht
- Narodowy Instytut Kardiologii Stefana Kardynała Wyszyńskiego Państwowy Instytut Badawczy, Warsaw, Poland
- United Kingdom (7):
  - Basildon & Thurrock University Hospitals (Essex CTC), Basildon
  - Health and Social Care Trust, Belfast
  - The Royal Bournemouth & Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - UH Bristol NHS Trust, Bristol Heart Institute, Bristol
  - Golden Jubilee National Hospital, Glasgow
  - St George's University Hospitals NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Wythenshawe Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Winter RW, Hoek R, Walsh SJ, Hanratty CG, Sprengers RW, Twisk JWR, Vegting I, Schumacher SP, Bom MJ, Verouden NJ, Henriques JP, Wilgenhof A, Viscusi MM, Teeuwen K, Opolski MP, Wolny R, Agostoni P, van Kuijk JP, Scholzel BE, Kraaijeveld AO, van Geuns RM, Dirksen MT, Heestermans AACM, Dens J, Bennett J, Haine SEF, Delewi R, Nap A, Spratt JC, Knaapen P; PROCTOR Trial Investigators. PCI of Native Coronary Artery vs Saphenous Vein Graft After Prior Bypass Surgery: A Multicenter, Randomized Trial. J Am Coll Cardiol. 2026 Jan 27;87(3):269-282. doi: 10.1016/j.jacc.2025.09.1577. Epub 2025 Oct 28. PMID 41159978